CLINICAL TRIAL: NCT06532357
Title: Evaluation of Satisfaction With Rimegepant and Triptans Utilizing Migraine Buddy Retrospective Data
Brief Title: A Study to Learn About the Benefit of Rimegepant Versus Triptans in Migraine Buddy App Users.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4951073; NCT06532357 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: acute treatment of migraine; rimegepant, triptans; Migraine Buddy App Users
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect information of the US users from the Migraine Buddy app between 20 October 2023 and 20 May 2024. Patients who used Nurtec and/or triptans as an acute treatment for migraine, with or without a background of preventive treatment (anti-CGRP, Botox or oral migraine preventive medications) and completed a survey were eligible for this study. Acute treatment is a short-term treatment. The aim of this retrospective analysis was to learn about the user´s satisfaction with Nurtec or the triptan. The level of satisfaction with Nurtec will be compared to the level of satisfaction with triptans. The benefit of this study is the real-life setting of the information collected. This means that the users were using the Migraine Buddy app for tracking their migraines in real life.

DETAILED DESCRIPTION:
This study will utilize retrospective data collected with the Migraine Buddy Mobile application to evaluate satisfaction of treatment with rimegepant and triptans. The study population for this study is Migraine Buddy users in the US who answered a survey about their acute treatments, displayed on the home page of the app. It generates reports that users can share with their doctors to help them establish a diagnosis and/or optimize treatment. For this retrospective study, only questions related to treatment satisfaction will be analyzed.

Users complete the satisfaction questions only once for each current acute migraine treatment. If a patient is using more than one acute treatment, they will be able to complete satisfaction questions for each acute treatment. Approximately two-thirds of the app users are currently using both rimegepant and triptans to acutely treat their migraine attacks. Questions are worded such that they ask specifically about the acute treatment e.g., Nurtec. For the surveys used in the 7-month time frame of this retrospective study, feasibility assessment showed that participants answered the satisfaction questions for a specific acute medication only once, in 97% of the cases. For the few users who responded to 2 or more waves of identical surveys, the most recent answer will be used for the analysis.

Data was gathered between October 20, 2023 & May 20, 2024, from users of the Migraine Buddy app through the "diary tracking" and the satisfaction questions were administered via survey and via the interactive data collection tool named "Taylor". All the data will be extracted from the Aptar Digital Health (ADH) platform existing database to perform the analysis described in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients who used Nurtec and/or triptans as an acute treatment for migraine, with or without a background of preventive treatment (anti-CGRP, Botox or oral migraine preventive medications).
* Male or female participants with migraine
* Having consented to the anonymous use of their data for research
* Currently using Nurtec and/or triptans to treat migraine attacks

Exclusion Criteria:

* Users who did not report using either medication for which they complete the survey within 60 days prior to the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: US users of the Migraine Buddy App who use rimegepant or triptans to treat their acute migraine attacks.
Sampling Method: Non-Probability Sample
Enrollment: 1536 (Actual)
Dates: Start 2024-06-09 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4951073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study, data was gathered between 30 October 2023 to 20 May 2024 from users of the Migraine Buddy application in the US who answered a survey about their acute treatments (rimegepant, or triptans) for migraine, displayed on the home page of the application. For the purpose of this retrospective study, only questions related to treatment satisfaction were analyzed.
Pre-assignment Details: As pre-specified, only variables/data collected were the self-reported satisfaction of Migraine Buddy users via a questionnaire accessible from the home screen of the application. Users completed the satisfaction questions only once for each current acute migraine treatment. A total of 1536 participants were enrolled in this study who completed the survey. There were few participants who were not exclusive and completed survey for both rimegepant and triptans.
Groups:
- Rimegepant: This arm included participants who used Migraine buddy application and answered the survey about satisfaction with rimegepant. No intervention was administered in this study.
- Triptans: This arm included participants who used Migraine buddy application and answered the survey about satisfaction with Triptans. No intervention was administered in this study.
Period: Period 1: Rimegepant User Survey
Arm/Group | Rimegepant | Triptans
Started | 708 | 0
Completed | 708 | 0
Not Completed | 0 | 0
Period: Period 2: Triptans User Survey
Arm/Group | Rimegepant | Triptans
Started | 0 | 845
Completed | 0 | 845
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For this retrospective study, as planned the only variables collected are the self-reported treatment satisfaction of Migraine Buddy users via a questionnaire accessible from the home screen of the application. Hence, Baseline data was not retrieved and not collected to be reported in the results.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rimegepant | Triptans | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized [unit: Participants] — Due to nature of study and retrieval of specific data/variables as planned, no age data was assessed and reported. Hence, Number Analyzed is 0.
Sex/Gender, Customized [unit: Participants] — Due to nature of study and retrieval of specific data/variables as planned, no sex/gender data was assessed and reported. Hence, Number Analyzed is 0.
Race and Ethnicity Not Collected [unit: participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction of Pain Intensity
Description: Participants responded about satisfaction with treatment for pain intensity using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment.
Time Frame: Up to 60 days post last usage of treatment (from retrospective data collection period of 7 months); available retrospective data was evaluated in this observational study of a single day
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 708 | 845
Participants
  Satisfied | 539 | 625
  Neutral | 130 | 178
  Dissatisfied | 39 | 42

2. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction With of Attack Duration
Description: Participants responded about satisfaction with of attack duration using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 708 | 845
Participants
  Satisfied | 524 | 571
  Neutral | 145 | 222
  Dissatisfied | 39 | 52

3. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction With Speed of Action
Description: Participants responded about satisfaction with speed of action using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 708 | 845
Participants
  Satisfied | 506 | 524
  Neutral | 154 | 272
  Dissatisfied | 48 | 49

4. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction With Migraine-Induced Cognitive Impact
Description: Participants responded about satisfaction with migraine-Induced cognitive impact using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 708 | 845
Participants
  Satisfied | 430 | 384
  Neutral | 237 | 377
  Dissatisfied | 41 | 84

5. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction With Relief of Other Symptoms
Description: Participants responded about satisfaction with relief of other symptoms using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment. Other symptoms included following parameters: photophobia, phonophobia, nausea, vomiting, sensitivity to light/sound/odors).
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 708 | 845
Participants
  Satisfied | 418 | 478
  Neutral | 243 | 301
  Dissatisfied | 47 | 66

6. Primary Outcome: Number of Participants Classified as Per Responses for Satisfaction of Tolerability
Description: Participants responded about satisfaction of tolerability using following responses: extremely satisfied, satisfied, slightly satisfied, neither satisfied nor dissatisfied, slightly dissatisfied, dissatisfied, extremely dissatisfied. Based on participants responses, the respondents were grouped into those who were satisfied (reported extremely satisfied/ satisfied/ slightly satisfied), neutral (reported neither satisfied nor dissatisfied) or dissatisfied (reported slightly dissatisfied/ dissatisfied/ extremely dissatisfied) with the treatment.
Time Frame: as for outcome 1
Population: Analysis population included all eligible participants whose data were retrieved and observed in the study. Here "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Rimegepant | Triptans
Number analyzed (Participants) | 447 | 845
Participants
  Satisfied | 385 | 554
  Neutral | 50 | 229
  Dissatisfied | 12 | 62

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events and all-cause mortality were not planned to be assessed/monitored during this study
Description: This observational retrospective data that existed as structured data by the time of study start. In these data sources, individual participant data were not retrieved or validated. The minimum criteria for reporting an adverse event (AE) (identifiable participant, identifiable reporter, a suspect product and event) was not met. Hence, AE were not assessed/evaluated which explains "0" participants at risk.
Arm/Group | Rimegepant | Triptans
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
For this retrospective study, the only variables collected are the self-reported satisfaction of Migraine Buddy users via a questionnaire accessible from the home screen of the app. Hence, Baseline data was not retrieved and is not presented in the study. As pre-specified, for the purpose of this retrospective study, only questions related to treatment satisfaction were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT06532357/Prot_SAP_000.pdf